CLINICAL TRIAL: NCT03721900
Title: A Phase 1 Pharmacokinetics and Pharmacodynamics of Ketamine Transdermal Drug Delivery System in Subjects With Sub-Optimally Responsive Major Depressive Disorders
Brief Title: Ketamine for Major Depressive Disorder
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shenox Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: SHX-C301
Record Dates: First submitted 2018-10-18; First posted 2018-10-26 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Major Depressive Disorder
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Each subject will receive one of the following: placebo, 20 mg (low dose), or 40 mg (high dose). All subjects will receive doses in the same order during 3 study periods
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SHX-001 Active Low Dose (Experimental): Ketamine transdermal patch
  Interventions: Drug: SHX-001 Active low dose
- Placebo (Placebo Comparator): placebo transdermal patch
  Interventions: Drug: Placebo
- SHX-001 Active high dose (Experimental): ketamine transdermal patch
  Interventions: Drug: SHX-001 Active High dose

INTERVENTIONS:
Drug: SHX-001 Active low dose — ketamine transdermal patch
  Other Names: Ketamine transdermal patch
  Arms: SHX-001 Active Low Dose
Drug: Placebo — transdermal patch
  Other Names: placebo transdermal patch
  Arms: Placebo
Drug: SHX-001 Active High dose — ketamine transdermal patch
  Other Names: ketamine transdermal patch
  Arms: SHX-001 Active high dose

SUMMARY:
The purpose of this study is to measure the amount of ketamine in blood over time in subjects diagnosed with Major Depressive Disorder (MDD) and explore the anti-depressive effects of ketamine delivered by transdermal patch.

DETAILED DESCRIPTION:
SHX-C301 is a Phase 1, first in human, single-blind, multi-center clinical study to evaluate the pharmacokinetics (PK), safety and antidepressant effects of SHX-001 transdermal patch low dose delivered based on prediction and high dose delivered based on the estimation from the low dose PK in subjects with MDD and sub-optimally controlled by standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Present a current depressive episode of at least 8 weeks
* Have a body mass index (BMI) of 18-35 kg/m2 (inclusive) at screening
* Agree to use adequate methods of contraception during the study (and for X days after discharge)

Exclusion Criteria:

* A history of alcohol consumption exceeding 14 drinks/week within the 5 years before study entry.
* Use of prescription or non-prescription drugs, vitamins, or dietary supplements within 14 days prior to the first dose of study medication except ongoing stable dose of antidepressant.
* Treatment with any investigational drug, use of any known CYP3A4 enzyme-inducing/inhibiting agents (e.g., barbiturates, phenothiazines, cimetidine, St. John's Wort) or herbal supplements within 7 days prior to the first dose of study medication
* A history of drug abuse or dependence within 180 days of screening
* A febrile illness within 5 days prior to the first dose of study medication.
* A known hypersensitivity to ketamine
* A history of use ketamine for Major Depressive Disorder and did not respond to ketamine
* Recent use of ketamine in any formulation for any indication (within 4 weeks prior to screening)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2018-12-28 (Actual); Primary Completion 2019-06-06 (Estimated); Study Completion 2019-06-06 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics of SHX-001 (Cmax) | 1 week
  Maximum observed plasma concentration
Pharmacokinetics of SHX-001 (Tmax) | 1 week
  Time of maximum observed plasma concentration
Pharmacokinetics of SHX-001 (T1/2) | 1 week
  Apparent terminal half-life

SECONDARY OUTCOMES:
Anti-depressive effects of SHX-001 | 1 week
  Antidepressant effects will be explored by assessing changes in depression assessments (clinician and self-rated)

OTHER OUTCOMES:
Safety objective as measured by Adverse Events (Safety and Tolerability of SHX-001) | Up to 10 weeks
  The safety and tolerability of SHX-001 transdermal patch as an adjunctive therapy to standard of care will be evaluated in subjects with MDD who are sub-optimally responsive to approved antidepressant.

CONTACTS AND LOCATIONS:
Overall Officials: Mason Freeman, MD, Study Director — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Clinical Research Site, Gaithersburg, Maryland
  - Clinical Research Site, Boston, Massachusetts
  - Clinical Research Site, Dayton, Ohio

IPD SHARING:
Plan to Share IPD: No